CLINICAL TRIAL: NCT03980301
Title: Screening Hepatitis Positive Women for Congenital Anomalies During Pregnancy and Assessment of Liver Status of Women
Brief Title: Screening Hepatitis Positive Women for Congenital Anomalies
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: hepatitis
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — screening of pregnant women with hepatitis c virus received treatment in first trimester for congenital anomalies

SUMMARY:
Hepatitis C virus is one of the virulent viruses

DETAILED DESCRIPTION:
Hepatitius positive women should be screened for congenital anomalies

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with hepatitis C virus received treatment during first trimester

Exclusion Criteria:

* pregnant women with hepatitis C virus who didnot receive treatment during first trimester

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women with hepatitis C virus
Study Population: Pregnant women with hepatitis C virus received treatment during first trimester
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
the number of pregnant women who will be diagnosed to have fetuses with congenital anomalies | within 6 months
  the number of pregnant women who will be diagnosed to have fetuses with congenital anomalies by us

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Study Chair — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt